CLINICAL TRIAL: NCT00425841
Title: Lokal Fortgeschrittenes Pankreas-Karzinom: Stereotaktische Radiotherapie Gefolfgt Von Gemox-Chemotherapie
Brief Title: Stereotactic Radiation Therapy and Combination Chemotherapy in Treating Patients Undergoing Surgery for Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000515934; KRDI-TUM-STRATEGIE-STR-242-LOR; EU-20659
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage III pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiosurgery

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Radiation: hypofractionated radiation therapy
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Drugs used in chemotherapy, such as gemcitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving stereotactic radiation therapy together with combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving combination chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving stereotactic radiation therapy together with combination chemotherapy works in treating patients undergoing surgery for locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response rate in patients undergoing surgery for locally advanced pancreatic cancer treated with stereotactic radiotherapy, gemcitabine hydrochloride, and oxaliplatin.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the time to disease progression in patients treated with this regimen.
* Determine the time to death in patients treated with this regimen.
* Determine perioperative morbidity and mortality in patients treated with this regimen.
* Determine the rate of R0 resections in patients treated with this regimen.
* Determine the histologic response rate in these patients.

OUTLINE:

* Neoadjuvant therapy: Patients undergo hypofractionated, stereotactic radiotherapy on days 1-5. Patients also receive gemcitabine hydrochloride IV over 100 minutes on day 1 and oxaliplatin IV over 120 minutes on day 2. Treatment with gemcitabine hydrocloride and oxaliplatin repeats every 2 weeks for 3 courses.
* Surgery: Patients with resectable disease undergo tumor resection. Patients with unresectable disease undergo a second course of neoadjuvant chemoradiotherapy followed by resection.
* Adjuvant therapy: Beginning 3-4 weeks after surgery, patients receive 3 more courses of chemotherapy as in neoadjuvant therapy.

After completion of study treatment, patients are followed every 3 months for up to 2 years.

PROJECTED ACCRUAL: A total of 29 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas or intrapancreatic bile duct carcinoma

  * Overall view of image morphology and CA19-9 (< 500 U/L) demonstrating pancreatic cancer allowed if histologic/cytologic confirmation is unavailable
* Locally advanced disease, meeting 1 of the following criteria:

  * Uncertain R0 resectability dependant on relation to portal vein, sinus confluens, superior mesenteric artery, and superior mesenteric vein (e.g., contact with portal vein, superior mesenteric vein, or arterial vessels, but < 180° encasement)
  * Unresectable pancreatic cancer (e.g., contact with portal vein, superior mesenteric artery or arterial vessels, > 180° encasement)
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 1 cm by spiral CT scan or MRI

  * Patients with no measurable disease may be assessed for feasibility only
* No distant metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 80-100%
* WBC ≥ 3,000/mm³
* Granulocyte count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine clearance > 30 mL/min
* Bilirubin ≤ 3.0 times upper limit of normal
* AST and ALT ≤ 2.5 times normal
* Alkaline phosphatase ≤ 2.5 times normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No secondary malignancy within the past 5 years that was not curatively treated
* No known intolerance to any of the study drugs
* No preexisting polyneuropathy > grade 1
* No active uncontrolled infection
* No cardiac insufficiency despite optimal medication
* No New York Heart Association class III or IV congestive heart failure
* LVEF ≥ 50% OR shortening fraction ≥ 25%
* No angina pectoris (at rest or under stress) unexplained by interventional cardiology within the past 6 months
* No myocardial infarction within the past 6 months
* No uncontrolled diabetes mellitus
* No other existing serious medical impairments that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No prior radiotherapy to the abdomen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2006-05; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Clinical response rate as assessed by RECIST criteria

SECONDARY OUTCOMES:
Toxicity as assessed by NCI-CTC criteria
Time to progression
Time to death
Perioperative morbidity and mortality
Rate of R0 resections
Histologic response rate

CONTACTS AND LOCATIONS:
Overall Officials: Florian Lordick, MD, Study Chair — Technical University of Munich
Locations (1):
- Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich, Germany